CLINICAL TRIAL: NCT01616368
Title: The Effects of Mindfulness Training on Eating Behaviors and Food Intake
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Principal Investigator, David Kearney, Staff Physician, Seattle Institute for Biomedical and Clinical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRB 00458
Record Dates: First submitted 2012-06-06; First posted 2012-06-11 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Obesity; Feeding Behavior
MeSH Terms: conditions — Obesity; Feeding Behavior | interventions — Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEAL (Experimental): Participation in an 8-week mindful eating course
  Interventions: Behavioral: Mindful Eating and Living Course

INTERVENTIONS:
Behavioral: Mindful Eating and Living Course — An eight week course designed to teach mindfulness skills with an emphasis on mindful eating.
  Other Names: MEAL

SUMMARY:
The investigators propose to study the effect of mindfulness training on the eating behaviors and dietary intake of overweight or obese persons. Mindfulness skills training involves bringing non-judgmental attention to thoughts, emotions and bodily sensations - including hunger and satiety cues. It is hypothesized that as subjects advance through the 8-week class series, developing their capacity for mindfulness and in effect learn to pay attention to the sensations, assumptions, cognitions, and beliefs that underlie their eating behaviors, that their eating behaviors will improve. Specifically, the investigators hypothesize that 1) there will be significant improvements in the areas of uncontrolled and emotional eating, 2) there will be significant decreases in total caloric intake and significant increases in fruits and vegetables, and 3) there will be a positive significant relationship between the frequency/consistency of mindfulness practice and improvements from baseline to follow-up measures.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) > 26

Exclusion Criteria:

* Psychotic disorders
* Poorly controlled bipolar disorder
* Borderline or antisocial personality disorder
* A diagnosed eating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in Eating behaviors | baseline, 2 months, 5 months
  The TFEQ will be administered. Subscales for emotional eating, uncontrolled eating and cognitive restraint will be assessed

SECONDARY OUTCOMES:
Change in Nutrition intake | baseline, 2 months, 5 months
  The ASA-24 and the DHQ will be administered to assess nutritional intake

CONTACTS AND LOCATIONS:
Overall Officials: David Kearney, MD, Principal Investigator — Seattle Institute for Biomedical and Clinical Research